CLINICAL TRIAL: NCT03684070
Title: Together we Move: A Multi-component Intervention to Increase Physical Activity for Ethnic Minority Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: Brandeis University (Other); Northeastern University (Other)
Responsible Party: Principal Investigator, Carina Katigbak, Assistant Professor, Boston College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19.001.01
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Physical Activity; Sedentary Lifestyle
Keywords: Older adults; Asian Americans; Chinese; behavior change
MeSH Terms: conditions — Motor Activity; Sedentary Behavior | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Walking (Experimental): FitBit + Lifestyle counseling/education session(8 weeks) + WeChat motivational messages and peer interaction
  Interventions: Behavioral: Self-Monitoring, peer support and motivational prompts
- Walking Only (Active Comparator): FitBit + Lifestyle counseling/education session(8 weeks)
  Interventions: Behavioral: Self-monitoring

INTERVENTIONS:
Behavioral: Self-Monitoring, peer support and motivational prompts — The intervention compares the effect of technologically delivered motivational messages, and peer support upon daily step counts.
  Arms: Enhanced Walking
Behavioral: Self-monitoring — Self-monitoring of data from wearable step count tracker
  Arms: Walking Only

SUMMARY:
The benefits of physical activity (PA) for healthy aging are well known; however < 16% of U.S. older adults meet the federal recommendations for moderate to vigorous PA (MVPA). Asian Americans (AA) are a fast-growing segment of the older adult U.S. population and are likely to have limited English proficiency, lower-incomes, and low PA levels. Older AA adults are under represented in clinical trials and as a result, evidence-based PA programs remain inaccessible. Similarly, while the number of PA interventions for older adults incorporating technology to promote and sustain behavior change is increasing, the applicability and efficacy of these approaches for AA is poorly understood. Thus, there is a critical need to develop and test innovative PA interventions for this at-risk group.

The primary objective of this study is to evaluate if a culturally and linguistically adapted community-based walking program enhanced with a cognitive behavioral intervention delivered via WeChat - a widely used Chinese social networking application - (enhanced walking) improves physical activity compared with walking only. Secondary objectives are to identify participant experiences in engaging in this platform to improve PA, and gain insights into the scalability of the intervention for future pivotal trials. The proposed research is a randomized, controlled trial that will recruit 60 community-dwelling Chinese older adults. The primary outcomes are PA (measured by FitBit step counts over time, and proportion meeting federal recommendations for moderate physical activity (MPA)). Secondary outcomes include patient-reported outcomes, and patient-reported experience measures. We aim to evaluate the acceptability of this enhanced program, and determine the feasibility of WeChat as a platform for increasing PA. The primary outcome will be analyzed using mixed effects ANOVA, and latent growth curve modeling. Secondary outcomes will be analyzed using linear regression. Semi-structured interviews will be conducted with participants upon program completion to identify contextual factors influencing application use, and thematic analysis will be used to examine relationships between these key factors.

Results from this study will provide information about the applicability of mobile technology in supporting PA improvement among older Chinese, and valuable insight on contextual factors influencing application effectiveness, which will inform the potential for adoption and scale.

DETAILED DESCRIPTION:
Implementation will be conducted at a single site, the Chinese Consolidated Benevolent Association of New England (CCA)). All subjects will consent to participate prior to continuing with study involvement as documented below.

Recruitment and Consent:

A convenience sample of a maximum of 60 participants (30 people per arm) will be recruited by placing ads in local newspapers, flyers at CBOs, local businesses, WeChat, and word of mouth. Interested individuals will call a dedicated voicemail box at Boston College and leave their contact information. A trained, bilingual member of the research team will contact interested individuals to obtain verbal consent for administration of the preliminary screening tool. If preliminary inclusion criteria are met, participants will be invited to an in-person secondary screening, where if deemed eligible to participate, signed informed consent for overall study participation will be obtained by a trained member of the study team in the participants' preferred language of communication (Mandarin or English). A $50 gift card will be offered to all enrolled participants.

Study methods:

Participation: After the consenting and initial (baseline) survey administration, assignment to the experimental or control group will be determined using a randomization list generated by a random number generator in R software. Both groups will meet on separate days and times to avoid contamination effects.

All participants will attend an orientation session to provide hands-on training on using the FitBit, and social networking platform (SNS) (as applicable).

A 2-week tech calibration period with one-on-one training with study staff will allow participants to acclimate to the FitBit, learn to use its features, and ask questions. Baseline FitBit data will be collected and monitored via Fitabase (a widely used and secure, research data management platform specific to FitBit data). This baseline data will allow the PI to generate an individualized walking prescription.

After this instructional trial period, all participants will be instructed to use the step-tracker's features to monitor their daily steps and progress towards meeting their individualized walking goals. All participants will attend 8 weekly educational sessions at the community center. Each day, those in the Enhanced Walking condition will receive 1-3 motivational messages related to physical activity and health; a monitoring protocol and database to document SNS interactions will be established. The Walking Only condition will not receive motivational messages through the SNS platform.

Surveys will be administered at study completion (8 weeks) and follow-up (12 weeks). FitBit data will be continually monitored throughout the study duration. A weekly adverse questionnaire will be administered by study staff in-person or via telephone when appropriate.

Follow-up outcomes: At the end of the study, participants from the experimental arm will be asked to attend a post-participation session where they will participate in a semi-structured interview to glean their experiences in using the SNS platform to promote physical activity.

Semi-structured interview questions will be posed to all clients who volunteer to participate in an interview session as part of the study. The interviews will be held at 4 weeks after the end of the study period. Interview questions and prompts were developed through a phenomenological lens to allow clients to elicit their own responses and experiences in the study. The interview guide will frame this discussion, and participant responses may be probed to gain further clarity or insight. The interviews will be audio recorded by study staff. Study staff will also write field notes to document client responses and other observations to supplement and provide context for the transcripts.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Chinese/Chinese American
* can communicate in Mandarin or English
* reside in Boston
* smartphone owners (iPhone or Android) with data plan
* no falls within last 6 months

Exclusion Criteria:

* + cognitive impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-18 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity | Through study completion, and average of 12 weeks
  Step counts as measured through FitBit tracker

SECONDARY OUTCOMES:
Self-efficacy for physical activity | Through study completion, and average of 12 weeks
  Self-Efficacy for Exercise (Resnick & Jenkins, 2000)
Qualitative Feedback | 4 weeks post-study completion
  Semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Carina Katigbak, PhD, Principal Investigator — Boston College
Locations (1):
- Boston College, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
All collected de-identified IPD will be shared within research consortium, but will not be available to external researchers.